CLINICAL TRIAL: NCT01516424
Title: A Randomized, Double-blinded, Double-dummy, Parallel-controlled and Multicenter Study to Investigate Blonanserin in Treatment of Schizophrenia When Compared With Risperidone
Brief Title: Efficiency Study to Investigate Blonanserin in Treatment of Schizophrenia When Compared With Risperidone
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sumitomo Pharma (Suzhou) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D4906011
Record Dates: First submitted 2012-01-18; First posted 2012-01-24 (Estimated); Results first posted 2018-11-26 (Actual); Last update posted 2018-11-27 (Actual); Status verified 2018-05

CONDITIONS: Schizophrenia
Keywords: Blonanserin
MeSH Terms: conditions — Schizophrenia | interventions — blonanserin; Risperidone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Blonanserin (Experimental): Antipsychotics
  Interventions: Drug: Blonanserin
- Risperidone (Active Comparator): Antipsychotics
  Interventions: Drug: Risperidone

INTERVENTIONS:
Drug: Blonanserin — Blonanserin tablets: 8 - 24mg/day; twice daily after breakfast and dinner; in the meantime, the placebo and positive drug were taken in whole tablets. When the morning and evening doses could not be administered equally, the evening dose should be greater than the morning dose. The interval between 2 dose escalations should not be shorter than 3 days.
  Other Names: Lonasen
  Arms: Blonanserin
Drug: Risperidone — Risperidone tablets: 2 - 6mg/day; twice daily after breakfast and dinner; in the meantime, the placebo and positive drug were taken in whole tablets. When the morning and evening doses could not be administered equally, the evening dose should be greater than the morning dose. The interval between 2 dose escalations should not be shorter than 3 days.
  Other Names: Risperdal
  Arms: Risperidone

SUMMARY:
A Randomized, Double-blinded, Double-dummy, Parallel-controlled and Multicenter Clinical trial to Investigate Blonanserin in Treatment of Schizophrenia when compared with Risperidone

DETAILED DESCRIPTION:
A Randomized, Double-blinded, Double-dummy, Parallel-controlled and Multicenter Clinical trial to Investigate Blonanserin in Treatment of Schizophrenia when compared with Risperidone

Trial drugs:

* Blonanserin group: Blonanserin tablets+Risperidone mimetic tablets
* Risperidone group: Risperidone tablets+Blonanserin mimetic tablets

Objectives of Study :

To evaluate the efficacy and safety of Blonanserin in treating schizophrenia

ELIGIBILITY:
Inclusion Criteria:

* Subject met Diagnostic and Statistical Manual of Mental Disorders(DSM)-IV-Text Revision(TR) criteria for a primary diagnosis of schizophrenia
* Patients are 18≤age<65 years of age on the day when informed consent is obtained.
* Subject had a PANSS total score ≥70 and 120≥ at Screening
* Subject had a score ≥4 on the PANSS at Screening and Baseline.
* Subjects are willing and able to comply with study protocol including treatment in hospital.
* Subjects or their legal guardians have signed the written informed consent form.

Exclusion Criteria:

* The subject was treatment with other Investigate product within 30 days.
* Subject had a history of treatment with long-acting drug for anti schizophrenia within 56 days.
* Subject had a history of treatment with clozapine within 28 days.
* Subject With parkinson disease,etc

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 267 (Actual)
Dates: Start 2012-02; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Niufan Gu, MD, Principal Investigator — Shanghai Mental Health Center
Locations (16):
- China (16):
  - Beijing Anding Hospital, Beijing, Beijing Municipality
  - Beijing Huilongguan Hospital, Beijing, Beijing Municipality
  - Peking University Sixth Hospital, Beijing, Beijing Municipality
  - Guangzhou Brain Hospital, Guangzhou, Guangdong
  - Hebei Province Mental Health Center, Baoding, Hebei
  - The First Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Henan Provincial Mental Hospital, Xinxiang, Henan
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Hunan Province Brain Hospital, Changsha, Hunan
  - Nanjing Brain Hospital, Nanjing, Jiangsu
  - Wuxi Mental Health Center, Wuxi, Jiangsu
  - Shanghai Mental Health Center, Shanghai, Shanghai Municipality
  - Xi'an Mental Health Center, Xi’an, Shanxi
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Tianjin Anding Hospital, Tianjin, Tianjin Municipality
  - First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan

RESULTS

PARTICIPANT FLOW:
Groups:
- Blonanserin: Blonanserin:
  Dosage Form: Tablet Dosage and Usage: 8~24mg/d ,b.i.d
- Risperidone: Risperidone:
  Dosage Form: Tablet Dosage and Usage: 2~6mg/d ,b.i.d
Period: Overall Study
Arm/Group | Blonanserin | Risperidone
Started | 131 (the patient number of randomization for Blonanserin Group) | 136 (the patient number of randomization for Risperidone Group)
Completed | 96 | 114
Not Completed | 35 | 22

BASELINE CHARACTERISTICS:
Population: 267 subjects in participant flow, 3 subjects randomized and not treated, 2 subjects does not have baseline PANSS scale, 1 subject take Blonanserin, which IWRS's indicate he should take Risperidone and no PANSS scale collectted after first dose. Those 6 subjects excluded from Baseline Population. The Baseline population have 261 subjects.
Groups:
- Blonanserin: Participants received 8-24mg tablet orally twice daily for 8 weeks
- Risperidone: Participants received 2-6mg tablet orally twice daily for 8 weeks
- Total: Total of all reporting groups
Arm/Group | Blonanserin | Risperidone | Total
Number analyzed (Participants) | 128 | 133 | 261
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 128 | 133 | 261
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 58 | 128
  Male | 58 | 75 | 133

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in PANSS(Positive and Negative Syndrome Scale) Total Score at Week 8
Description: Mean change in Positive and Negative Syndrome Scale total score from baseline to Week 8 at the end of treatment. PANSS is an interview-based measure of the severity of psychopathology in adults with psychotic disorders. It have 30 evaluation items, which include 7 positive sub-scale, 7 negative sub-scale and 16 general psychopathology sub-scale on a score of 1 to 7. The total score is the sum of the 30 scale items. The minimum score is 30 and the maximum score is 210. Patient with PANSS total scores<70 is the normal,but the scores>120 is more serious.Change=(Week 8 Score - Baseline score)
Time Frame: From baseline to the end of study、week 8(day 56)or before other antipsychotic taken.
Population: 267 subjects in participant flow, 3 subjects randomized and not treated, 2 subjects does not have baseline PANSS scale, 1 subject take Blonanserin, which randomized to Risperidone group and no PANSS scale collected after first dose. Those 6 subjects excluded from Baseline Population. The Baseline population have 261 subjects.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Blonanserin | Risperidone
Number analyzed (Participants) | 128 | 133
score on a scale
  ITT analysis: At the end of treatment | -30.59 (18.53) | -33.56 (16.89)
  PPS analysis: At the end of treatment: number analyzed (Participants) | 121 | 113
  PPS analysis: At the end of treatment | -33.71 (17.02) | -36.31 (14.09)
Statistical Analysis 1: Comparison: Blonanserin vs Risperidone; ANCOVA was employed to compare the changes of PANSS scores at week 8 relative to the baseline in these 2 groups. Least Squares Means for the differences in changes between the 2 groups (μ blonanserin - μ risperidone) and the two-sided 95% Confidence Interval were calculated in accordance with the main model. H0: Compared with risperidone, blonanserin reduced more than 7.0 in mean change in PANSS total score from baseline at week 8 of treatment (μ blonanserin-μ risperidone> 7.0); Test type: Non-Inferiority or Equivalence — The power is 80%, non-inferiority margin is 7.0; p < 0.05, ANCOVA — Satisfaction with the non-inferiority criteria was determined by the upper limit of confidence interval. If the upper limit of 95% confidence interval was less than 7.0, then non-inferiority was concluded; Study center and grouping as fixed effects; Mean Difference (Final Values) = 3.69, 95% CI 2-sided [-0.36 to 7.75] — This is ITT analysis data
Statistical Analysis 2: Comparison: Blonanserin vs Risperidone; ANCOVA was employed to compare the changes of PANSS total scores at end of treatment relative to the baseline in these 2 groups. LSMeans for the differences in changes between the 2 groups (μ blonanserin - μ risperidone) and the two-sided 95% Confidence Interval were calculated in accordance with the main model. H0: Compared with risperidone, blonanserin reduced more than 7.0 in mean change in PANSS total score from baseline at week 8 of treatment (μ blonanserin-μ risperidone> 7.0); Test type: Non-Inferiority or Equivalence — The power is 80%, non-inferiority margin is 7.0; p < 0.05, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Study center and grouping as fixed effects; Mean Difference (Final Values) = 2.94, 95% CI 2-sided [-0.76 to 6.65] — This is PPS analysis data

2. Secondary Outcome: Mean Change in PANSS Subscale Score at the End of Treatment
Description: Mean Change in PANSS subscale score at the end of treatment at 8 weeks the frame of 8 weeks is from baseline
Time Frame: week 8
Reporting Status: Not Posted

3. Secondary Outcome: Mean Change in PANSS 5-factor Model
Description: Mean change in PANSS 5-factor model from baseline at Week 8
Time Frame: Week 8
Reporting Status: Not Posted

4. Secondary Outcome: Mean Change in PANSS Symptom Scores
Description: Mean change in PANSS symptom scores from baseline at Week 8
Time Frame: Week 8
Reporting Status: Not Posted

5. Secondary Outcome: Mean Change in PANSS Symptom Scores From Baseline at Each Visit
Description: Mean change in PANSS symptom scores from baseline at each Visit from baseline at week 8
Time Frame: Each Visit
Reporting Status: Not Posted

ADVERSE EVENTS:
Description: Safety analysis set (SS, the primary analysis set for safety evaluation) SS of this study included all randomized subjects who have received at least 1 dose of the trial drug.
  The SS population have 130 subjects in Blonanserin group, 134 subjects in Risperidone group.
Arm/Group | Blonanserin | Risperidone
Serious Adverse Events (participants affected / at risk) | 1/130 | 3/134
Other Adverse Events (participants affected / at risk) | 126/130 | 122/134
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Blonanserin (N=130) | Risperidone (N=134)
chicken pox (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — One subject (random number 234) in blonanserin group developed "chicken pox" and recovered after quarantine, symptomatic and supportive treatment; in the investigator's opinions, this case was unrelated to the study drug.
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Gastrointestinal foreign matter (Gastrointestinal disorders) | 0 (0) | 1 (1)
fever of unknown origin (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Blonanserin (N=130) | Risperidone (N=134)
Palpitations (Cardiac disorders) | 8 (11) | 13 (15)
Tachycardia (Cardiac disorders) | 3 (4) | 5 (5)
Sinus bradycardia (Cardiac disorders) | 2 (2) | 5 (5)
Sinus arrhythmia (Cardiac disorders) | 2 (2) | 3 (3)
Sinus tachycardia (Cardiac disorders) | 2 (2) | 3 (4)
Galactorrhea (Endocrine disorders) | 0 (0) | 3 (3)
Blurred vision (Eye disorders) | 0 (0) | 3 (3)
constipation (Gastrointestinal disorders) | 21 (28) | 22 (34)
diarrhea (Gastrointestinal disorders) | 4 (5) | 4 (4)
Nausea (Gastrointestinal disorders) | 3 (6) | 5 (5)
Oropharyngeal pain (Gastrointestinal disorders) | 3 (3) | 4 (4)
Toothache (Gastrointestinal disorders) | 2 (3) | 4 (5)
Vomit (Gastrointestinal disorders) | 2 (2) | 3 (3)
Fatigue (Immune system disorders) | 3 (3) | 6 (7)
sleepiness (Immune system disorders) | 4 (4) | 0
Fever (Immune system disorders) | 0 (0) | 3 (3)
Abnormal liver function (Hepatobiliary disorders) | 9 (9) | 17 (17)
Nasopharyngitis (Infections and infestations) | 14 (16) | 20 (23)
Upperrespiratory tract infection (Infections and infestations) | 7 (8) | 4 (4)
Tinea pedis (Infections and infestations) | 3 (3) | 0 (0)
Serum prolactin increase (Investigations) | 68 (68) | 90 (90)
Alanine aminotransferase increase (Investigations) | 7 (7) | 8 (8)
Aspartate aminotransferase increase (Investigations) | 4 (4) | 5 (5)
Blood triglycerides increase (Investigations) | 3 (3) | 6 (6)
Lipid increase (Investigations) | 2 (2) | 5 (5)
Body weight increase (Investigations) | 2 (2) | 4 (4)
Blood cholesterol increase (Investigations) | 2 (2) | 3 (3)
Transaminase increase (Investigations) | 2 (2) | 3 (3)
Blood potassium decrease (Investigations) | 3 (3) | 1 (1)
Poor appetite (Metabolism and nutrition disorders) | 4 (5) | 3 (3)
Hyperlipidemina (Metabolism and nutrition disorders) | 3 (3) | 3 (3)
Extrapyramidal disorders (Nervous system disorders) | 63 (71) | 39 (41)
Dizziness (Nervous system disorders) | 5 (7) | 6 (7)
Tremor (Nervous system disorders) | 3 (3) | 2 (2)
Headache (Nervous system disorders) | 3 (3) | 1 (1)
Excitement (Psychiatric disorders) | 28 (32) | 16 (19)
Insomnia (Psychiatric disorders) | 24 (31) | 18 (25)
Anxiety (Psychiatric disorders) | 11 (11) | 11 (12)
Poor sleep quality (Psychiatric disorders) | 6 (6) | 6 (6)
Dysphoria (Psychiatric disorders) | 4 (4) | 2 (2)
Somnipathy (Psychiatric disorders) | 3 (3) | 4 (4)
Akathisia (Psychiatric disorders) | 4 (4) | 2 (2)
Diffculty falling asleep (Psychiatric disorders) | 3 (4) | 3 (3)
Irritability (Psychiatric disorders) | 4 (5) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 2 (2)
Stuffy nose (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (4)
Expectoration (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No